CLINICAL TRIAL: NCT01768611
Title: Association of Single Nucleotide Polymorphisms in the Gene Coding GLUT-1 and Diabetic Nephropathy in Brazilian Patients With Type 1 Diabetes Mellitus
Brief Title: SLC2A1 Variants and Diabetic Nephropathy
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FMUSP-LIM25-001
Record Dates: First submitted 2012-12-17; First posted 2013-01-15 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Nephropathy.
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Withou Diabetic Nephropathy: Patients who have persistent normoalbuminuria (<30 mg/g creatinine or <20 μg/min).
- Incipient Nephropathy: Patients who have persistent microalbuminuria (30-300 mg/g creatinine or 20-200 μg/min).
- Overt Diabetic Nephropathy: Patients who have persistent macroalbuminuria (>300 mg/g creatinine or >200 µg/min), proteinuria (>500 mg/24 h) or renal replacement therapy.

SUMMARY:
Cells damaged by hyperglycemia are unable to downregulate glucose entrance in presence of high extracellular glucose resulting in intracellular activation of deleterious biochemical pathways. Expression of GLUT-1, the major glucose transporter in mesangial cells, is increased and participates in the induction of diabetic nephropathy. Variants in the gene encoding GLUT-1 (SLC2A1) have been associated to this diabetic complication. The aim of this study was to test whether polymorphisms in SLC2A1 confer susceptibility to diabetic nephropathy in Brazilian type 1 diabetes patients.

DETAILED DESCRIPTION:
In this study, 449 patients, included between October 2004 and October 2012, were sorted into three groups according to diabetic nephropathy stages: without (persistent normoalbuminuria, n=248), incipient (microalbuminuria, n=82) and overt diabetic nephropathy (macroalbuminuria or proteinuria or renal replacement therapy, n=119). Measurements of urinary albumin-to-creatinine ratio (ACR) or urinary albumin excretion rate (UAER) were used to define DN: patients with persistent normoalbuminuria (<30 mg/g creatinine or <20 μg/min) were classified as without DN (n=248); patients presenting persistent microalbuminuria (30-300 mg/g creatinine or 20-200 μg/min) were classified as having incipient DN (n=82); and patients presenting persistent macroalbuminuria (>300 mg/g creatinine or >200 µg/min), proteinuria (>500 mg/24 h) or renal replacement therapy were classified as having overt DN (n=119). Genotyping of polymorphisms was performed by Real Time PCR using fluorescent -labelled probes.

ELIGIBILITY:
Inclusion Criteria:

* Overt 10 years of Diabetes Mellitus

Exclusion Criteria:

* Patients presenting autoimmune diseases, HIV or HCV infections
* Patients with glomerular filtration rate < 60 mL min-1 1.73 m2 without diabetic retinopathy

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 449 patients with type 1 diabetes (56.4% female, mean age 36.0±11.0 years) were included between October 2004 and October 2012. Inclusion criterion was type 1 diabetes duration ≥10 years. The patients presented a mixed ethnic background (European Caucasian, African, Amerindian and Asian of several different countries of origin), which reflects the Brazilian population.
Sampling Method: Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2004-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Plasmatic Creatinine | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Côrrea-Giannela, Doctor, Principal Investigator — Hospital Clínicas/Faculdade de Medicina da USP
Locations (1):
- Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil